CLINICAL TRIAL: NCT01358201
Title: Treatment Protocol For All Fragile Patients Ph' Negative Over 55 Years
Brief Title: PETHEMA LAL-07FRAIL: All Treatment In Fragile Patients Ph' Negative Over 55 Years
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PETHEMA LAL-07FRAIL
Record Dates: First submitted 2011-05-18; First posted 2011-05-23 (Estimated); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Vincristine; Dexamethasone; Methotrexate; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: vINCRISTINE
Drug: Dexamethasone
Drug: Methotrexate
Drug: Cytosine arabinoside

SUMMARY:
The biological characteristics of the adult LAL, karyotypic and phenotypic particular, are fundamentally different from those of Acute Lymphoblastic Leukemia (ALL) children and, consequently, the results of treatment are substantially lower. Additionally, elderly patients tolerate the drugs considered relatively low-key in the management of the LAL and suffer more toxicity. Although the LAL is much more common in patients over 60 years of age than in younger adults, older adults with ALL are clearly underrepresented in prospective controlled studies. A good portion of elderly patients are not able to tolerate the intensity of the standard treatment applied to children or young adults and a significant portion of them receive only palliative or supportive treatment. The data in the literature relating specifically to the elderly population are scarce and most of them have obtained a stratification by age of study designed for young people (CALGB, GMALL, PETHEMA). To date, the group's recommendation was to treat PETHEMA the LAL-96RI protocol for elderly patients because this protocol less aggressive than those used in high-risk ALL. However, the development of inhibitors of tyrosine kinases LAL effective in Bcr / abl positive, a relatively common type of LAL in the older patient, requires a differentiated treat these patients. Moreover, analysis of data from patients treated so far with the LAL-96RI protocol has shown mediocre results even for LAL Bcr / abl negative. This analysis also showed a significant benefit in survival related to the reduction of treatment (removal of the L-asparaginase during induction and cyclophosphamide at the end of induction) attributed to a reduction in toxicity

DETAILED DESCRIPTION:
Prephase (days -5 to -1) Dexamethasone 10 mg/m2 bolus day EV for 5 days (-5 to -1). Supplementary treatment: hydration minimum 2000 ml / day. allopurinol 300 mg / day. gastric protection (as center). daily monitoring of blood glucose daily monitoring of renal function.

Intrathecal treatment (diagnosis and prophylactic / therapeutic) day -5: 12 mg were administered intrathecal methotrexate. The morphological study of the CSF will be defining initial CNS involvement by LAL. Although it is recommended immunophenotypic study of CSF, the definition of CNS involvement by LAL (and its therapeutic consequences) based on morphological observation of blasts in CSF cytocentrifuge.

Remission induction :

Tolerance prephase period can be used to establish the final indication of treatment (standard protocol or frail patients). Day 0 is free of treatment and is considered as +1 the first day of induction.

Systemic treatment

* Vincristine (VCR) 1 mg (absolute dose) EV 1, 8, 15 and 22.
* Dexamethasone (DEX): 10 mg/m2 EV, IM or PO days 1-2, 8-9 days 15-16, 22-23.

Intrathecal chemotherapy

Triple therapy was administered with methotrexate (MTX), cytosine arabinoside (ARA-C) and hydrocortisone, days 1, 8, 15 and 22 (five doses total prophylactic between prephase and induction):

MTX 12 mg ARA-C 40 mg Dexamethasone 4 mg

If initial infiltration of the CNS is administered once every 72 hours until the disappearance of blast cell morphology CSF (cytocentrifugation) in at least two consecutive taps. Alternatively be administered liposomal cytarabine (DepoCyt) fortnightly if authorized by the center or in the context of a clinical trial

Maintenance treatment of first year :

Maintenance during the first year will start after full recovery after induction and after complete reassessment of the disease (including myelogram) and will last until one year from the time of documentation of complete remission.

The basic treatment to include mercaptopurine 50 mg/m2 PO day and methotrexate 20 mg/m2 IM weekly.

Once every 3 months will be added to maintenance treatment a "mini-reinduction" consisting

* VCR: 1 mg (absolute dose), i.v., day 1.
* Dexamethasone 40 mg / day, i.v. or p.o., days 1-2.
* Not considered more doses of triple intrathecal therapy. Reinduction only be practiced during the first year after remission, so a total of 4 quarterly.

Maintenance of the second year:

After the first year of maintenance will perform a complete reassessment of the disease (including myelogram) and if the patient remains in complete remission maintenance will continue (without reinduction) until two years from the time of diagnosis.

The initial dose of mercaptopurine and methotrexate will be identical to the first year. Must comply (by increases or decreases of 20% of the dose) to maintain the numbers of neutrophil counts between 1.5 and 3x109/l and platelets above 100x109 / L

ELIGIBILITY:
Inclusion Criteria:

Adults over 55 years diagnosed with acute lymphoblastic leukemia Ph 'negative and not previously treated with frailty (> 3 points in the Charlson comorbidity index)

Exclusion Criteria:

LAL

1. L3 type mature B phenotype (sIg +) or cytogenetic abnormalities characteristic of Burkitt LAL (t [8, 14], t [2, 8], t [8, 22]).

2 . biphenotypic acute leukemias and bilinear 3 . acute undifferentiated leukemia 4 . Patients with a Charlson comorbidity index less than or equal to 3 (and therefore that could potentially benefit from more intensive treatment PETHEMA LAL-07OLD).

5 . General condition affected (grades 3 and 4 WHO scale), not attributable to the LAL.

6 . LAL Ph 'positive (though still must register their LAL07OPH specific protocol).

7 . Lack of consent by the patient to use their clinical data

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-05 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy in terms of response rate | 5 years

SECONDARY OUTCOMES:
Efficacy in terms disease free survival | 5 years
Efficacy in terms of global survival | 10 years

CONTACTS AND LOCATIONS:
Locations (73):
- Spain (73):
  - H. Son Llatzer, Palma de Mallorca, Balearic Islands
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Juan Canalejo, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Fundación Hospital Alcorcón, Alcorcón
  - Hospital de Alcorcón, Alcorcón
  - Hoapital General, Alicante
  - Hospital General de Alicante, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clinic y Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau., Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Valle Hebrón, Barcelona
  - Institut Català d'oncología, Barcelona
  - Basurtuko Ospitalea, Basurto
  - Hospital de Cruces, Bilbao
  - Complejo Hospitalario de Cáceres, Cáceres
  - Complejo Hospitalario Reina Sofía, Córdoba
  - Area Hospitalaria Juan Ramón Jimenez, Huelva
  - Hospital Médico Quirúrgico Ciudad de Jaén, Jaén
  - H. de Jerez, Jerez de la Frontera
  - Complejo Hospitalario León, León
  - Hospital Arnau de Vilanova, Lleida
  - Complexo Hospitalario Xeral-Calde, Lugo
  - Clínica La Concepción, Madrid
  - Clínica Puerta de Hierro, Madrid
  - Clínica Rúber, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital 12 de Octubre. Madrid, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid
  - Hospital de Fuenlabrada, Madrid
  - Hospital de la Princesa, Madrid
  - Hospital de Madrid, S.A.- Norte Hospital General, Madrid
  - Hospital La Paz, Madrid
  - Althaia, Xarxa Asistencial de Manresa, Manresa
  - Fundación Hospital Sant Joan de Déu de Martorell, Martorell
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Complejo Hospital Costa del Sol, Málaga
  - H. Carlos Haya, Málaga
  - Hospital Carlos Haya, Málaga
  - Hospital General Morales Meseguer, Murcia
  - Hospital Morales Messeguer. Murcia, Murcia
  - Hospital Sta. Maria del Rosell, Murcia
  - Hospital Central de Asturias, Oviedo
  - Hospital del Río Carrión, Palencia
  - Complejo Asistencial Son Dureta, Palma de Mallorca
  - Complejo Hospitalario de Pontevedra_Hospital Montecelo, Pontevedra
  - Complejo Hospitalario de Pontevedra_Hospital Provincial, Pontevedra
  - Corporació Sanitaria Parc Taulí, Sabadell
  - Hospital Clinico Universitario, Salamanca
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Clínica Sant Camil, Sant Pere de Ribes
  - Hoaspital Marqués de Valdecilla, Santander
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Complejo Hospitalario Regional Virgen del Rocío, Seville
  - Hospital Joan XXIII, Tarragona
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hoapital La Fe, Valencia
  - Hospital Clínico de Valencia., Valencia
  - Hospital Clínico de Valencia, Valencia
  - Hospital Clínic, Valencia
  - Hospital Dr Pesset, Valencia
  - Hospital General, Valencia
  - Hospital La Fe, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Complejo Hospitalario Universitario de Vigo, Vigo
  - Comarcal de Vinaros, Vinaròs
  - Hospital Clinico Lozano Blesa, Zaragoza
  - Hospital Lozano Blesa. Zaragoza, Zaragoza

REFERENCES:
- See also: Pethema Foundation — https://www.fundacionpethema.es/